CLINICAL TRIAL: NCT01410968
Title: A Feasibility and Safety Study of Vaccination With Poly-ICLC and Peptide-pulsed Dendritic Cells in Patients With Metastatic, Locally Advanced, Unresectable, or Recurrent Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carolyn Britten (Other)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Carolyn Britten, Chief, Hematology/Oncology Division, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101498
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccination (Experimental): vaccination with investigational Poly-ICLC & peptide-pulsed dendritic cells
  Interventions: Drug: vacc. w/ Poly-ICLC & peptide-pulsed dendritic cells

INTERVENTIONS:
Drug: vacc. w/ Poly-ICLC & peptide-pulsed dendritic cells — Intradermal injection of 1x107 peptide-pulsed dendritic cells followed by intramuscular injection of 30 micrograms per kilogram Poly-ICLC on days 0, 14, 28 and 42. Additional dose of 30 micrograms per kilogram Poly-ICLC on days 3, 17, 31 and 45. Treatment given via one 56-day cycle. Leukapheresis performed at baseline for dendritic cell generation.

SUMMARY:
The purpose of this study is to provide a safety and feasibility basis for future studies addressing the hypothesis that subcutaneous vaccination with dendritic cells loaded with multiple antigenic epitopes expressed by pancreatic tumor in combination with systemic administration of Poly-ICLC (Hiltonol) will induce anti-tumor immunity.

DETAILED DESCRIPTION:
Primary Objectives

1. Assess the safety of this treatment by evaluating the qualitative and quantitative toxicities in this group of patients.
2. Determine the feasibility of generating dendritic cells and administering these cells as a vaccine to patients.

Secondary Objectives

1. Assess anti-tumor activity after vaccination, measured by change in tumor burden and overall survival.
2. Assess immunological responses after vaccination (antigen-specific T cell cytokine production, antigen-specific T cell frequencies by tetramer analysis, and DTH reactions)

ELIGIBILITY:
Eligibility Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma that is metastatic, locally advanced, unresectable, or recurrent. Patients with endocrine or neuroendocrine tumors, lymphoma of the pancreas, or ampullary cancer are not eligible. If the histologic diagnosis is based on a metastatic site, the histology must be compatible with pancreatic cancer.
* Patient must not have clinically significant ascites.
* Patients must be HLA-A2 positivity by serological testing.
* Prior surgery is allowed provided at least 14 days has elapsed between surgery and registration. Prior radiation/chemo is allowed provided that at least 28 days have elapsed since the last treatment.
* One or more tumors measurable on CT scan per RECIST 1.1. (Eisenhauer)
* Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* Age > 18 years.
* Patient must have an expected life expectancy greater than 3 months.
* Signed, written IRB-approved informed consent.
* A negative pregnancy test (if female).
* Acceptable organ function:
* Bilirubin < 3 times upper limit of normal (CTCAE Grade 2 baseline)
* AST (SGOT), ALT (SGPT) < 3 x ULN (CTCAE Grade 1 baseline)
* Serum creatinine < 1.5 XULN (CTCAE Grade 1 baseline)
* Acceptable hematologic status:
* Absolute neutrophil count > 1000 cells/mm3,
* Platelet count > 75,000 (plt/mm3), (CTCAE Grade 1 baseline)
* Hemoglobin > 9 g/dL.
* Urinalysis: No clinically significant abnormalities.
* PT and PTT < 1.5 X ULN after correction of nutritional deficiencies that may contribute to prolonged PT/PTT.
* No evidence of clinically significant, uncontrolled cardiovascular, endocrine, or infectious disease.

Exclusion Criteria

* Patients must not have any serious uncontrolled acute or chronic medical condition that would interfere with this treatment. An example would be an active acute or chronic infection requiring antibiotics
* Patients must not have significant ongoing cardiac problems, myocardial infarction within the last six months, uncontrolled hypertension, unstable angina, uncontrolled arrhythmia or congestive heart failure.
* Patients with known brain metastases are not eligible. However, brain-imaging studies are not required for eligibility if the patient has no neurologic signs or symptoms. If brain-imaging studies are performed, they must be negative for disease.
* Patients must have no plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol treatment.
* Due to the undetermined effect of this treatment regimen in patients with HIV-1 infection and the potential for serious interaction with anti-HIV medications, patients known to be infected with HIV are not eligible for this study.
* Due to the possibility of harm to a fetus or nursing infant from this treatment regimen, patients must not be pregnant or nursing. Women and men of reproductive potential must have agreed to use an effective contraceptive method.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 years
  Any protocol deviations will be described and the protocol schedule will be re-assessed to improve feasibility of implementation if necessary. The proportion of patients successfully completing the protocol (i.e., without deviations) will be reported with a one-sided 90% confidence interval. If the observed feasibility rate is >0.80, the lower limit will be no lower than 0.60.
Safety | 2 Years
  All toxicities will be reported by type and grade and tabulated. To provide a safety characterization of the treatment regimen, it is important that common toxicities be observed in this phase of study for planning the next phase of research.

SECONDARY OUTCOMES:
Efficacy | 2 years
  Graphical displays of tumor size (as a percentage of baseline) over time. A subject's best response (i.e., complete response, partial response, stable disease or progressive disease) will be reported. Time to disease progression from baseline for each patient will be reported. Time to death will be reported in the same manner. These results will be summarized using proportions with confidence intervals and Kaplan-Meier curves, although the confidence limits are expected to be wide based on the small sample size.
Immunological Responses | 2 years
  Antigen-specific T cell frequencies, antigen-specific T cell cytokine production and DTH reactions will be assessed.
  For T cell-based functional analysis, each measurement will be performed with the three peptides telomerase, CEA, and survivin. Transformation of the continuous outcomes will be logged. Post measurements will be normalized by the baseline value (i.e. we will subtract the baseline value from each of the post vaccination measurements after the log transformations). Each of these measures will be displayed graphically over time for each patient to observe modulations in these measures. If appropriate based on the distribution of values over time, linear longitudinal regression will be used to model the change in these outcomes over time. Appropriateness will be based on the consistency of trends across patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Mehrotra S, Britten CD, Chin S, Garrett-Mayer E, Cloud CA, Li M, Scurti G, Salem ML, Nelson MH, Thomas MB, Paulos CM, Salazar AM, Nishimura MI, Rubinstein MP, Li Z, Cole DJ. Vaccination with poly(IC:LC) and peptide-pulsed autologous dendritic cells in patients with pancreatic cancer. J Hematol Oncol. 2017 Apr 7;10(1):82. doi: 10.1186/s13045-017-0459-2. PMID 28388966